CLINICAL TRIAL: NCT01272479
Title: Comparison of Prohepcidin, Inflammation and Iron Homeostasis in Hemodialysis Patients With and Without Chronic Hepatitis C
Brief Title: Prohepcidin, Inflammation and Iron Homeostasis in Hemodialysis Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Istanbul University Scientific Research Projects, Istanbul University
Other Study IDs: 1692
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2009-11

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Hepatitis C
Keywords: hemodialysis; hepatitis C; inflammation; iron stores; prohepcidin
MeSH Terms: conditions — Hepatitis C; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- HCV (+): Hemodialysis patients with chronic hepatitis C
- HCV (-): Hemodialysis patients without chronic hepatitis C
- Control: Healthy volunteers

SUMMARY:
The aim of this study is to address questions regarding the link among hepcidin, hematological iron markers, inflammation and hepatitis C in HD patients. In attempt to address this issue, we planned to measure serum levels of hepcidin prohormone (pro-hepcidin), inflammatory and iron parameters.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is the most common cause of chronic liver disease in the world and also common among chronic hemodialysis (HD) patients. Patients with chronic HCV often have increased liver iron, a condition associated with reduced sustained response to antiviral therapy, more rapid progression to cirrhosis, and development of hepatocellular carcinoma; however, little is known about the mechanism of iron accumulation in the liver. Recently identified hepcidin, a 25-amino acid peptide hormone exclusively synthesized in the liver, is thought to be a key regulator for iron homeostasis and is induced by infection and inflammation. Hepcidin expression is modulated by iron stores, so that it decreases in iron deficiency to facilitate iron absorption while it increases in iron repletion to prevent pathological overload. Interleukin (IL)-6 has been proposed as a major inducer of hepcidin, via direct transcriptional activation of hepatic hepcidin expression by binding to its receptor complex containing gp130 to activate janus kinase (JAK) and activator of transcription 3 (STAT 3).

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients

Exclusion Criteria:

* Patients positive for hepatitis B virus surface antigen (HBsAg)
* Patients previously diagnosed nonrenal cause of anemia other than iron deficiency
* Patients with an evidence of active or occult bleeding
* Patients received blood transfusion within the past 4 months
* Patients with a history of malignancy, end-stage liver disease, or chronic hypoxia
* Patients with a history of recent hospitalization or infection requiring antibiotics within the past 4 weeks.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients on chronic hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Association of prohepcidin and inflammation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Caliskan, Principal Investigator — MD
Locations (1):
- Division of Nephrology, Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Nemeth E, Tuttle MS, Powelson J, Vaughn MB, Donovan A, Ward DM, Ganz T, Kaplan J. Hepcidin regulates cellular iron efflux by binding to ferroportin and inducing its internalization. Science. 2004 Dec 17;306(5704):2090-3. doi: 10.1126/science.1104742. Epub 2004 Oct 28. PMID 15514116